CLINICAL TRIAL: NCT06970197
Title: Effect of Simulation and Out-of-Class Educational Activities Intervention on Sustainability in Nursing Students: A Randomized Controlled Trial
Brief Title: The Effect of Simulation and Out-of-Class Educational Activities on Sustainability Among Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ummuhan Okur, Lecturer, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 85
Record Dates: First submitted 2025-04-13; First posted 2025-05-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sustainability; Randomized Controlled Trial; Public Health Nursing
Keywords: nursing; sustainability; simulation; out-of-class education

STUDY DESIGN:
Intervention Model Description: This research is a parallel group pre-test-post-test randomized controlled experimental design.
Who Masked: Outcomes Assessor
Masking Description: Since the researcher was the person who monitored the implementation of the intervention to the students in the intervention group and actively carried out the process, researcher blinding could not be applied. However, blinding will be applied by ensuring that the data collection tools are made by a faculty member who is not involved in the research. In order to prevent bias in the evaluation of the data, statistical blinding will be applied by ensuring that the statistics of the data collected as a result of the research are made by an independent statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The control group will not receive any intervention and will attend other courses within the scope of their undergraduate education. After the intervention part of the study is completed, the educational content given to the intervention group will be shared with the control group.
- simulation group (Experimental): After the theoretical training, the students in the simulation group will participate in three different simulation applications for three weeks. The simulation application will be carried out using high-fidelity simulation (standard patient and simulator) in the simulation unit and will include prebriefing, simulation application and debriefing sessions.
  Interventions: Other: simülation group
- out-of-class educational activities group (Experimental): Three out-of-class educational activities were planned by the researchers within the scope of experiential learning.
  Interventions: Other: out-of-class educational activities group

INTERVENTIONS:
Other: simülation group — İncludes high reality simulation applications.
  Arms: simulation group
Other: out-of-class educational activities group — It includes a tour of the sales facility, a sapling planting activity and an "action for the environment" activity to provide experiential learning.
  Arms: out-of-class educational activities group

SUMMARY:
This research will be conducted to evaluate the effects of simulation and out-of-class education activities intervention given to students using the Ecological Planet Health Model on environmental literacy, sustainability knowledge, sustainability attitudes in nursing and sustainable consumption behaviors of nursing students. The research will be conducted at Selçuk University Faculty of Nursing and Selçuk University Selçuk Pharmacy Simulation Unit located in Konya province. The study group consists of second-year students (n=204) studying and attending courses at Selçuk University Faculty of Nursing in the Spring Semester of 2024-2025 Academic Year. The sample size was determined as a total of 72 students.

DETAILED DESCRIPTION:
This study includes two intervention groups (Intervention 1: Simulation Group, Intervention 2: Out-of-Class Educational Activities Group). Both groups received joint theoretical training on climate change and sustainability in the same classroom for seven weeks. A follow-up test was administered in the eighth week, and then, according to the random assignment determined at the beginning of the study, Intervention Group 1 (24 students) participated in simulation applications for three weeks, while Intervention Group 2 (24 students) participated in out-of-class educational activities for three weeks. The preparation of SWOT analyses and action plans for both groups will be determined. These courses are expected to be prepared and submitted within three weeks. The training program will be integrated into the 14-week Climate Sustainability and Sustainability curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Being a second year undergraduate nursing student

Exclusion Criteria:

* Working in any health institution or organization,
* Being a member of any environmental institution or organization,
* Being a foreign student

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Sustainability awareness scale knowledge dimension | 14 weeks
Sustainability attitudes in nursing survey | 14 weeks
Sustainable consumption behavior scale | 14 weeks
Environmental literacy scale | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personally, I don't prefer this situation.

REFERENCES:
- [Background] Richardson J, Heidenreich T, Alvarez-Nieto C, Fasseur F, Grose J, Huss N, Huynen M, Lopez-Medina IM, Schweizer A. Including sustainability issues in nurse education: A comparative study of first year student nurses' attitudes in four European countries. Nurse Educ Today. 2016 Feb;37:15-20. doi: 10.1016/j.nedt.2015.11.005. Epub 2015 Nov 10. PMID 26646207
- [Background] Richardson J, Grose J, Bradbury M, Kelsey J. Developing awareness of sustainability in nursing and midwifery using a scenario-based approach: Evidence from a pre and post educational intervention study. Nurse Educ Today. 2017 Jul;54:51-55. doi: 10.1016/j.nedt.2017.04.022. Epub 2017 Apr 29. PMID 28477563
- [Background] Abhijith K, Kumar P, Gallagher J, McNabola A, Baldauf R, Pilla F, Broderick B, Di Sabatino S, Pulvirenti B, 2017. Air pollution abatement performances of green infrastructure in open road and built-up street canyon environments-A review. Atmospheric environment, 162, 71-86.